CLINICAL TRIAL: NCT00940303
Title: An Open Label, Single-arm, Phase II Study to Evaluate the Efficacy and the Feasibility of Bevacizumab (Avastin) Based on a FOLFOXIRI Regimen Until Progression in Patients With Previously Untreated Metastatic Colorectal Carcinoma(OPAL-Study)
Brief Title: OPAL Study: A Study of Avastin (Bevacizumab) in Combination With FOLFOXIRI in Patients With Previously Untreated Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20514; 2008-001180-11
Record Dates: First submitted 2009-07-06; First posted 2009-07-16 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Bevacizumab; Irinotecan; Leucovorin; Oxaliplatin

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: 5-FU; Drug: bevacizumab [Avastin]; Drug: irinotecan; Drug: leucovorin; Drug: oxaliplatin

INTERVENTIONS:
Drug: 5-FU — 3200mg/m2 continuous iv infusions, day 1 every 2 weeks
Drug: bevacizumab [Avastin] — 5mg/kg iv infusion, day 1 every 2 weeks
Drug: irinotecan — 165mg/m2 iv infusion, day 1 every 2 weeks
Drug: leucovorin — 200mg/m2 iv infusion, day 1 every 2 weeks
Drug: oxaliplatin — 85mg/m2 iv infusion, day 1 every 2 weeks

SUMMARY:
This single arm study will assess progression-free survival, feasibility of use and safety of Avastin in combination with 5-FU/FA, oxaliplatin and irinotecan (FOLFOXIRI) as first line treatment in patients with metastatic colorectal cancer. Patients will receive up to 12 bi-weekly cycles of Avastin (5mg/kg iv) in combination with this standard neoadjuvant chemotherapy regimen followed by up to 40 bi-weekly cycles with Avastin plus 5-FU/FA. The anticipated time on study treatment is until disease progression, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-70 years of age;
* metastatic colorectal cancer scheduled for standard first line chemotherapy;
* at least 1 measurable lesion;
* ECOG performance score of 0 or 1.

Exclusion Criteria:

* prior chemotherapy for metastatic colorectal cancer;
* prior (neo)adjuvant chemotherapy/radiotherapy of a non-metastatic malignancy completed within 6 months prior to study entry;
* concomitant malignancies other CRC;
* history or evidence of CNS disease unrelated to cancer.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2009-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | assessed every 8 weeks up to week 102, 3-monthly during follow-up

SECONDARY OUTCOMES:
Overall survival; proportion of patients achieving R0 resectability; objective response rate (complete response [CR] and partial response [PR]); proportion of patients completing 12 cycles of chemotherapy. | assessed every 4 weeks up to week 102 and at the end of follow-up period
Proportion of patients with NCI-CTC grade 3-5 adverse events; adverse events, laboratory parameters, ECOG performance status. | Throughout study, laboratory analyses every 2 weeks, ECOG assessment every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (13):
- Germany (13):
  - Berlin
  - Bochum
  - Celle
  - Dessau
  - Freiburg im Breisgau
  - Fulda
  - Hamburg
  - Hanover
  - Leer
  - Magdeburg
  - Nuremberg
  - Stade
  - Villingen-Schwenningen

REFERENCES:
- [Derived] Stein A, Atanackovic D, Hildebrandt B, Stubs P, Brugger W, Hapke G, Steffens CC, Illerhaus G, Bluemner E, Stohlmacher J, Bokemeyer C. Upfront FOLFOXIRI+bevacizumab followed by fluoropyrimidin and bevacizumab maintenance in patients with molecularly unselected metastatic colorectal cancer. Br J Cancer. 2015 Sep 15;113(6):872-7. doi: 10.1038/bjc.2015.299. Epub 2015 Sep 3. PMID 26335608